CLINICAL TRIAL: NCT00918177
Title: Dual Release Gastric Retentive AP09004, Vs. Active Control; a Pharmacokinetic/Pharmacodynamic, Comparative, Safety Evaluation in Parkinson's Patients
Brief Title: An Evaluation of the Pharmacokinetics and Pharmacodynamics of AP09004 in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intec Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN 09 004
Record Dates: First submitted 2009-06-01; First posted 2009-06-11 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2010-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early patients (Experimental)
  Interventions: Drug: AP09004; Drug: Carbidopa/Levodopa, immediate release
- Moderate Patients (Experimental)
  Interventions: Drug: AP09004; Drug: Carbidopa/Levodopa, immediate release

INTERVENTIONS:
Drug: AP09004
Drug: Carbidopa/Levodopa, immediate release

SUMMARY:
The purpose of this study is to evaluate blood level profiles of multiple oral doses of AP09004 vs. active control and to determine its safety and efficacy in Parkinson's patients.

ELIGIBILITY:
* Subjects between the ages of 18 and 75 years of age inclusive;
* For early patients only: Subject with Parkinson's disease with a stable response to Levodopa (not suffering from "wearing off") and currently treated with IR-Carbidopa/Levodopa containing 300-500mg Levodopa per day up to 4 doses per day.
* For group 3 only: Subject with Parkinson's disease experiencing predictable motor fluctuations, end of dose "wearing off", defined by the patient's report of at least two episodes daily of a decline in function from peak benefit, with at least 2-3 hours OFF a day at the discretion of the PI (does not include early morning akinesia). Only patients with end of dose wearing off for at least 3 months will be included.
* For moderate patients only: patients who are currently treated with IR-Carbidopa/Levodopa containing 600-900mg Levodopa, in divided dose, per day.
* Subject has been stable at current CD/LD dose for at least 1 months
* Hoehn and Yahr stages I-III
* If subject is taking dopamine agonists, the dose has been stable for at least 1 month
* Other then Parkinson's disease, the subject is in satisfactory health, as assessed by physical examination, blood test (biochemistry and hematology). No abnormality on clinical examination and blood tests that in the opinion of the Physician responsible will compromise safety or interfere with study procedures.

Exclusion Criteria:

* Subjects who have participated in another clinical trial within the last 30 days;
* Subjects with atypical Parkinsonism
* Subject has significant history of cardiac, pulmonary, hepatic or renal disease or other condition or any major complication/illness which, in the opinion of the physician responsible, contraindicates his/her participation.
* Subject with symptomatic gastroparesis with frequent vomiting (at least once a week).
* Subjects with a history of clinically defined GERD, peptic ulcer or any gastrointestinal surgery other than appendectomy or herniotomy, or with any gastrointestinal disorder likely to influence drug absorption, or with any history of inflammatory bowel disease, irritable bowel syndrome, severe gastrointestinal narrowing, or frequent nausea or emesis, regardless of etiology.
* Prior gastro-intestinal surgery or current gastrointestinal conditions of clinical significance including ulcers, diarrhea, vomiting, bleeding, intestinal obstruction or inflammatory bowel disease, which, in the opinion of the physician responsible, contraindicates his/her participation.
* History of drug or alcohol abuse.
* Subject has a history of allergy to any component of the dosage form or any other allergy, which, in the opinion of the physician responsible, contraindicates his/her participation.
* Subjects suffering from psychological disorders that in the opinion of the physician responsible may interfere with full participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate blood level profiles and safety of the AP09004

SECONDARY OUTCOMES:
Efficacy of AP09004 on motor scores in Parkinson's patients

CONTACTS AND LOCATIONS:
Overall Officials: T Gurevich, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; R. Djaldetti, Prof. MD, Principal Investigator — Rabin Medical Center; O. Cohen, MD, Principal Investigator — Sheba Medical Center; Ilana Schlesinger Schlesinger, MD, Principal Investigator — Rambam Health Care Campus, Haifa, Movement Disorders and Parkinson's Disease; Ron Milo, M.D, Principal Investigator — Barzilai Medical Center, Department of Neurology, Movement disorders unit, Ashkelon, Israel; Peter Farkas, M.D, Principal Investigator — Department of Neurology, Clalit University Medical Center; Marieta Anca-Herschkovitsch, M.D, Principal Investigator — Edith Wolfson , Dept. of Neurology, Movement Disorders Unit.
Locations (7):
- Israel (7):
  - Barzilai Medical Center, Department of Neurology, Movement disorders unit,, Ashkelon
  - Department of Neurology, Clalit University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa, Movement Disorders and Parkinson's Disease, Haifa
  - Edith Wolfson , Dept. of Neurology, Movement Disorders Unit., Holon
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - TASMC, Tel Aviv